CLINICAL TRIAL: NCT04707261
Title: A Prospective, Randomized, Double-blind, Multicenter Study on the Association Between Dapagliflozin-induced Improvement and Anemia in Heart Failure Patients (ADIDAS)
Brief Title: Association Between Dapagliflozin-induced Improvement and Anemia in Heart Failure Patients (ADIDAS)
Acronym: ADIDAS
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Xiangtan Central Hospital (Other)
Collaborators: Second Xiangya Hospital of Central South University (Other); ZhuZhou Central Hospital (Other)
Responsible Party: Principal Investigator, Jianping Zeng, President of Xiangtan Centeral Hospital, Xiangtan Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020/12/01
Record Dates: First submitted 2020-12-31; First posted 2021-01-13 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Anemia; Heart Failure
Keywords: Heart Failure; Anemia; Dapagliflozin
MeSH Terms: conditions — Anemia; Heart Failure | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dapagliflozin (Experimental): Dapagliflozin with standard-of-care therapies for heart failure, including sacubitril/valsartan or ACEI/ARB, beta-blocker, MRA, ICD and CRT
  Interventions: Drug: Dapagliflozin
- Placebo (Placebo Comparator): Standard-of-care therapies for heart failure, including sacubitril/valsartan or ACEI/ARB, beta-blocker, MRA, ICD and CRT
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin — Participants will receive dapagliflozin 10 mg once daily
  Other Names: FORXIGA
  Arms: Dapagliflozin
Drug: Placebo — Participants will receive placebo 10 mg once daily
  Arms: Placebo

SUMMARY:
The primary objective of this study is to investigate the hemoglobin change and association between hemoglobin change and readmissions due to heart failure, and all-cause death in patients with heart failure treated with dapagliflozin or placebo.

DETAILED DESCRIPTION:
Study Description Brief Summary: The primary objective of this study is to investigate the hemoglobin change and association between hemoglobin change and readmissions due to heart failure, and all-cause death in patients with heart failure treated with dapagliflozin or placebo.

Detailed Description: Heart failure is one of the most serious health concerns in the world, and it also remains the most common reason for hospitalization in older individuals. In patients with heart failure, anemia is associated with an increased risk of hospitalization and all-cause mortality. The DAPA-HF trial demonstrated that dapagliflozin was able to reduce the risk of worsening heart failure (HF) events and cardiovascular death comparing to placebo in patients with reduced ejection fraction on top of standard of care.

This is an investigator-initiated, interventional, prospective, double-blind study. The primary objective is to investigate whether anemia correction is one of the prerequisites and determinants related to the beneficial effects of dapagliflozin in patients with heart failure. Impact of dapagliflozin treatment on hemoglobin level, heart failure-related readmission and all-cause death will be observed in comparison with placebo in heart failure patients receiving guideline recommended standard therapy during the 3months, 6 months and 1 year follow up.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between the ages of 18 and 100 years.
2. Elevated NT-proBNP or BNP levels on admission.
3. Ejection fraction of 50% or less, and New York Heart Association (NYHA) class II, III, or IV symptoms.

Exclusion Criteria:

1. Treatment with SGLT2-i during the past 3 months of admission,or previous intolerance of an SGLT2 inhibitor.
2. Severe (eGFR <30 mL/min/1.73 m^2 by CKD-EPI), unstable or rapidly progressing renal disease at the time of randomization.
3. Pregnant or breast feeding female patients.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1990 (Estimated)
Dates: Start 2021-08-06 (Actual); Primary Completion 2025-05-05 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Composite number of hospital admissions for Heart Failure (HF) and all-cause death | 1 year
  Total number of deaths and heart failure hospitalizations in one year

SECONDARY OUTCOMES:
Change in the Kansas City Cardiomyopathy Questionnaire (KCCQ) score | Baselin, 3 months, 6 months, and 1 year
  The Kansas City Cardiomyopathy Questionnaire (KCCQ) is a 23-item, self-administered instrument that quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life. Scores are transformed to a range of 0-100, in which higher scores reflect better health status.
Change in 6-minute walk distance (6MWD) | Baselin, 3 months, 6 months, and 1 year
  This test measures the distance that a patient can quickly walk on a flat, hard surface in a period of 6 minutes.
Change in hemoglobin | Baselin, 3 months, 6 months, and 1 year
  g/L

CONTACTS AND LOCATIONS:
Overall Officials: Jianping Zeng, Ph.D., Study Chair — Xiangtan Central Hospital; Shenghua Zhou, Ph.D., Study Director — Second Xiangya Hospital of Central South University; Chengming Wang, Ph.D., Study Director — ZhuZhou Central Hospital; Fanghua Xu, M.D., Study Director — The First People's Hospital of Xiangtan City; Zhiqiang Cai, M.D., Study Director — Xiangtan People's Hospital; Chonglun Zhou, M.D., Study Director — Xiangxiang People's Hospital
Locations (1):
- Xiangtan Central Hospital, Xiangtan, Hunan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zeng J, Zhu Y, Zhao W, Wu M, Huang H, Huang H, Wu C, Zhou X, Zhou S, Wang C, Yin K, Xu F, Cai Z, Li X, Cheng H, Xie Y, Tan Z, Hu X, Liao D, Wang Y. Rationale and Design of the ADIDAS Study: Association Between Dapagliflozin-Induced Improvement and Anemia in Heart Failure Patients. Cardiovasc Drugs Ther. 2022 Jun;36(3):505-509. doi: 10.1007/s10557-021-07176-0. Epub 2021 Mar 29. PMID 33779938